CLINICAL TRIAL: NCT05464368
Title: Comparison of 18F-RO948, 18F-MK6240, and 18F-GTP1 Radiopharmaceuticals in Patients With Alzheimer Disease and Older Controls
Brief Title: R21 Roche: 3-Way Tau Tracers in AD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 202204181
Record Dates: First submitted 2022-06-23; First posted 2022-07-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — (18F)GTP1

STUDY DESIGN:
Intervention Model Description: Cohort 1Summary: BBBM/Amyloid PET scan A+;CDR .5 or1,Inclusive;arterial lines(N=8) Cohort 2Summary:BBBM/Amyloid PET scan A-;CDR 0;arterial lines; (N=8) Cohort3 Roche Supplement Summary: BBBM/Amyloid PET scan A+; CDR 0,.5 and/or 1(approx. 1/3rdof participants in each CDR score); can shorten total scan time or add break(N=22)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: (A+; CDR = .5, 1; AD) (Experimental): Unblinded and randomized to receive either 18F-RO948or 18F-MK6240 for PET Scan #1. PET scan #2 will be either 18F-RO948or 18F-MK6240 NOT received in PET scan #1. If a 3rdPET scanoccurs,this third scanwill always be [18F]GTP1.
  Interventions: Drug: [18F]RO-948; Drug: 18F-MK6240; Drug: 18F-GTP1
- Cohort 2: (A-; CDR=0; OC) (Experimental): Unblinded and randomized to receive either 18F-RO948or 18F-MK6240 for PET Scan #1. PET scan #2 will be either 18F-RO948or 18F-MK6240 NOT received in PET scan#1.If a 3rdPET scan occurs, this third scan will always be [18F]GTP1.
  Interventions: Drug: [18F]RO-948; Drug: 18F-MK6240; Drug: 18F-GTP1
- Cohort 3: (A+; CDR = 0, .5, 1; AD) (Experimental): Unblinded and randomized to receive 18F-RO948or 18F-MK6240 or [18F]GTP1for PET Scan #1. PET scan #2 will be 18F-RO948or 18F-MK6240 or [18F]GTP1NOT received in PET scan #1. PET scan # 3 will be 18F-RO948or 18F-MK6240 or [18F]GTP1NOT received in PET scan #1 or #2. Efforts will be made to include about 1/3 CDR = 0; 1/3 CDR = .5; 1/3 CDR = 1 in Cohort 3. Efforts will also be made to completethe study with about equal numbers of subjects whose PET scan #1 start with each of the three tracers.
  Interventions: Drug: [18F]RO-948; Drug: 18F-MK6240; Drug: 18F-GTP1

INTERVENTIONS:
Drug: [18F]RO-948 — Johns Hopkins University has conducted the first in human study in collaboration with Roche for 18F-RO948and found that 18F-RO948isa promising radioligand for imaging tau pathology in AD, showing excellent brain uptake and displaying little off-target binding(22, 17, 34).The injected activity for18F-RO948will be as low as practicable, while still allowing accurate quantification of the PET images.The injected dose of 370MBq(10mCi)has been selected based on the radiation dose estimates for18F-RO948gathered in human subjects provided by Michael Stabin, Ph.D., and in accordance with the principle that radiation doses should be "as low as reasonably achievable".
  This radiotracer will be manufactured on site in the Mallinckrodt Institute of Radiology Cyclotron Facility, a certified Nuclear Pharmacy.
Drug: 18F-MK6240 — 18F-MK6240 is an investigational PET radiotracer discovered by Merck Research Laboratories and is being developed by Cerveau Technologies, Inc.,for imaging neurofibrillary tangles (NFTs)in the brains of people withAlzheimerdisease.18F-MK6240 has been reported to exhibit good kinetics with high binding levels to brain regions associated with deposition of neurofibrillary tangles in people with AD(35,36).The tracer has been used to monitor the progression of AD.The injected activity for18F-MK6240 will be as low as practicable, while still allowing accurate quantification of the PET images.The injected dose will be 185MBq(5mCi) has been selected based on the radiation dose estimates gathered in human subjects(37)and in accordance with the principle that radiation doses should be "as low as reasonably achievable."
  This radiotracer will be manufactured on site in the Mallinckrodt Institute of Radiology Cyclotron Facility, a certified Nuclear Pharmacy.
Drug: 18F-GTP1 — 18F-GTP1is anInvestigational tau PET radiotracer being developed by Genentech for imaging intraneuronal neurofibrillary tangles in patients with AlzheimerDisease. 18F-GTP1 has been reported to exhibit high affinity and selectively for tau pathology, favorable dosimetry and brain kinetics. Degree of 18F-GTP1-specific binding increased withAD severity, could differentiate diagnostic cohorts, and monitor longitudinal change in tau burden.
  18F-GTP1 will be provided from LMI sourced through Illinois or New Jersey certified location.

SUMMARY:
This is an open label study to compare three new generation TAU radioligands, 18F-RO948 (formerly known as 18F-6958948), 18F-MK6240, and [18F]GTP1for imaging of taupathy and demonstrate their absence of off-target binding in patients with Alzheimer disease (AD) and older healthy controls (OC). The study will directly compare AD and OC with these three next-generation TAU radioligands and compare each of them with historical data of the current most widely used first generation radioligand, 18F-AV1451. Upto38 (30 AD (Amyloid +)and 8 OC (Amyloid -), matched for age and sex with A+ subjects) male and female subjects aged 50-100 will be enrolled in this study protocol: up to 8 for Cohort 1, up to 8 for Cohort 2, and up to 22 for Cohort 3. The study consists of three cohorts: Cohort 1: Up to8 AD subjects (A+; CDR 0.5 and 1)will receive two PET scans in random order, with receiving either18F-RO948 or18F-MK6240 at the first scan. A third scan with 18F-GTP1is possible, depending on timing and radiotracer availability Cohort 2:Up to8 OC (A-; CDR=0)subjects will receive two PET scans in random order, with receiving either18F-RO948or 18F-MK6240 at the first scan. A third scan with 18F-GTP1is possible, depending on timing and radiotracer availability Cohort 3:Up to 22 (A+; CDR = 0, .5 and 1) subjects will receive three PET scans in random order, with receiving 18F-RO94818F-MK6240 or18F-GTP1at the first scan. Efforts will be made to include about 1/3 CDR = 0, 1/3 CDR .5, and 1/3 CDR 1 in Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 50 to 100 years of age: Female subjects must be either surgically sterile or post-menopausal for at least 1 year or, Women of child bearing potential must commit to use a barrier contraception method for the duration of the study in addition to either an intra uterine device or hormonal contraception started at least 1 month prior to the first dose of radiotracer and until follow-up. Male subjects and their partners of childbearing potential must agree to use an effective method of contraception and will not donate sperm during the study. Barrier method must include use of a spermicide.
* Subjects who sign an IRB approved informed consent prior to any study procedures. Subjects deemed incapable of informed consent must have informed consent provided by a legally authorized representative. For AD subjects, capacity for consent will be determined using the Alzheimer Disease Research Center's questions
* Subjects who in the opinion of the investigator based on medical history and physical exam can tolerate the PET scan procedures,and can safely tolerate tracer administration and the scanning procedures.
* If subjects are on any concomitant medication, the indication and dosage of these medicines should be stable for at least 4 weeks prior to study start with the expectation that no relevant changes in use or dose will occur throughout the trial.
* Body mass index BMI between 18 and 32 kg per m2, Body weight less than 300 pounds
* Older Controls must have normal cognitive function, including a normal CDR = 0 as judged by the investigator for OC.
* AD subjects must have a diagnosis of probable AD, according to the National Institute of Neurological and Communicative Disorders and Stroke Alzheime rDisease and Related Disorders Association criteria with a CDR >0 to 1 and positive CSF or amyloid PET Scan.
* AD subjects must have a reliable person able to accompany the subject to all visits and answer questions about the subject.
* AD subjects must have a positive florbetapiro, amyloid blood-based biomarkers(BB BM), or amyloid-beta and tau CSF levels, which in the opinion of the principal investigator is consistent with a diagnosis of AD.

Exclusion Criteria:

* History or presence of a neurological diagnosis other than AD that may influence the outcome or analysis of the scan results; examples include but are not limited to stroke, traumatic brain injury, space occupying lesions, non-Alzheimer tauopathies, and Parkinson's disease.
* Subjects with a medical history that includes known autosomal dominant AD mutations in amyloid precursor protein APP or presenilin PS1, PS2 or mutations in genes that cause other types of autosomal dominant familial dementia, e.g., tau MAPT
* History or presence of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal, metabolic, endocrine, or CNS disease or other medical conditions that are not well controlled, may put the subject at risk, could interfere with the objectives of the study, or make the subject unsuitable for participation in the study for any other reason in the opinion of the principal investigator.
* Clinically relevant pathological findings in physical examination, ECG, or laboratory values at the screening assessment that could interfere with the objectives of the study.
* Known history of clinically significant infectious disease including AIDS or serological indication of acute or chronic hepatitis B or C or HIV infection.
* Women of childbearing potential must not be pregnant, or nursing and serum human chorionic gonadotropin HCG must be negative at the time of Screening Visit, and urine HCG must be negative on all subsequent visits.
* Loss or donation of more than 450 mL blood in the 4 months before screening or donation of plasma within 14days of screening or history of bleeding disorder or presence of anticoagulants
* Current symptoms of allergy and or severe allergy to drugs in medical history.
* History of drug or alcohol abuse or positive result from urine screen for drugs of abuse. AD subjects on prescribed narcotics medications will not be excluded if urine drug screen is positive for the documented narcotic drugs.
* Have received an investigational medication within the last 3 months or 5 elimination half-life, whichever is longer, prior to administration of the radiotracer.
* Has had or is planning to have exposure to ionizing radiation that in combination with the study related tracer administrations and scanning procedures would result in a cumulative exposure that exceeds 5.0 rem over a 12-month period of time.
* Contraindications of previous or study screening MRI
* History of, or suffers from, claustrophobia or feels that he or she will be unable to lie still on their back in the MRI or PET scanner.
* Subjects with hearing impairment, illiteracy, non-English speakers, or English as a second-language (since there is no direct medical benefit to participants).
* Subjects who have not completed at least 2 COVID-19 vaccination injections.16. Subjects who will not wear mask over nose and mouth during all visits except

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Amyloid positivity of patients with Alzheimer disease or positive memory or thinking problem CDR assessment compared to amyloid negative older healthy controls. | 37-44 days
  Amyloid positivity will be measured by either PET or CSF or blood-based biomarker (BBBM). Investigators will analyze the correlation between image quality and amyloid positivity to support any conclusions that will determine if 18F-MK6240 or 18F-RO948 has better discrimination between Amyloid + and Amyloid - subjects.
Imaging capability of 18F-RO948, 18F-MK6240 and 18F-GTP1 in patients with Alzheimer disease or positive memory or thinking problem CDR assessment, and amyloid negative older healthy controls, as compared to 18F-AV1451. | 37-44 days
  Using 18F-RO948, 18F-MK6240, and [18F]GTP1 for imaging of taupathy in patients with Alzheimer's disease (AD) and older healthy controls (OC), investigators will directly compare images and amyloid positivity (Outcome 1) of AD and OC to determine discrimination ability. Investigators will compare all images and amyloid positivity of AD and OC to data gathered using 18F-AV1451 to determine if the new radiotracers are able to outperform this well-known tracer.
Correlation between imaging capability of 18F-RO948, 18F-MK6240 and 18F-GTP1 and amyloid positivity of patients with Alzheimer disease or positive memory or thinking problem CDR assessment compared to amyloid negative older healthy controls. | 37-44 days
  Investigators will compare the quality of images to the previously measured amyloid positivity to support any conclusions that will determine if 18F-MK6240 or 18F-RO948 has better discrimination between Amyloid + and Amyloid - subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Dean F Wong, Principal Investigator — Head Researcher/Professor of Radiology
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Share information with NIH according to guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code